CLINICAL TRIAL: NCT00326612
Title: Intranasal Midazolam Versus Rectal Diazepam for the Home Treatment of Seizure Activity in Pediatric Patients With Epilepsy
Brief Title: Intranasal Midazolam Versus Rectal Diazepam for Treatment of Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Primary Children's Hospital (Other)
Responsible Party: Principal Investigator, Maija Holsti, Associate Professor Division of Pediatric Emergency Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15275
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-09

CONDITIONS: Seizures
Keywords: Seizures
MeSH Terms: conditions — Seizures | interventions — Midazolam; Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Midazolam 0.2mg/kg (Active Comparator): GIve once for seizure longer than 5 minutes
  Interventions: Drug: Midazolam
- Rectal Diazepam 0.3-0.5 mg/kg (Active Comparator): Given once for seizure longer than 5 minutes
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Midazolam — Intranasal Midazolam 0.2 mg/kg given once for seizures longer than 5 minutes.
  Other Names: Diastat
  Arms: Intranasal Midazolam 0.2mg/kg
Drug: Diazepam — Rectal Diazepam (Diastat) given once for seizure greater than 5 minutes.
  Other Names: Versed
  Arms: Rectal Diazepam 0.3-0.5 mg/kg

SUMMARY:
The investigators will conduct a randomized controlled trial comparing the use of nasal midazolam, using a Mucosal Atomization Devise, to rectal diazepam for the treatment of acute seizure activity in children under the age of 18 years with epilepsy in the community setting. The primary hypothesis is that nasal midazolam will be more effective and have shorter seizure time compared to rectal diazepam in the community. The secondary hypotheses are that patients treated with nasal midazolam will have fewer respiratory complications, emergency department visits, and admissions.

DETAILED DESCRIPTION:
Study Design: This is a prospective randomized controlled study.

Study Procedures: Parents/guardians will be provided with a stopwatch to help record seizure times on the "Parent Form". All parents of children who have a seizure lasting longer than five minutes will be randomized to treat their seizure with the study medication (either rectal diazepam or nasal midazolam). If a parent treats a child with a study medication for seizure activity they are required to call "911". Families will be instructed to only give one dose of the study medication. If the seizure persists, EMS may give a second medication and transport the patient to the ED as per their established protocol. All parents/guardians who participate in this study will be asked to fill out a "Pre-study Form" (to be filled out during enrollment into the study) and a "Parent Form" for every seizure that is treated with the study medication. They will be given a stamped returned envelope to return the questionnaire. Once the study medication is used once, they will be done with the study. Any further need of home rescue medications to treat acute seizure activity will be coordinated by their neurologist. If questions arise, a study coordinator will be available by phone. In addition, parents/guardians will be contacted by phone every two months and questioned at clinic visits to audit compliance of reporting of seizures/hospitalizations, adverse events and answer any questions that arise. The study packet also instructs all families to call the study coordinator immediately if any expected or unexpected complication occurs. The study coordinator will be called on all ED visits and hospitalizations. We will then collect and analyze adverse events to compare them between the two groups. Any ER visit or hospitalization will be considered an adverse event and will be analyzed for its relationship to the seizure or medication. All adverse events will be reported to the IRB. See Table 1 for doses for the two study medications.

ELIGIBILITY:
Inclusion Criteria:

* Children seventeen years and under will be identified through a Pediatric Neurology clinic at Primary Children's Medical Center,
* Known seizure disorder, AND
* Either have or will be prescribed a rescue anti-epileptic (rectal diazepam, or Diastat) for home use by their neurologist.

Exclusion Criteria:

* The neurologist does not prescribe a rescue medication for home use,
* 18 years of age or older,
* They have absence seizures, OR
* They have been prescribed lorazepam for home use for seizure activity.

Ages: 1 Week to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 358 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maija Holsti, MD, MPH, Principal Investigator — University of Utah; Francis Filloux, MD, Study Chair — University of Utah; Jeff Schunk, MD, Study Chair — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Harbord MG, Kyrkou NE, Kyrkou MR, Kay D, Coulthard KP. Use of intranasal midazolam to treat acute seizures in paediatric community settings. J Paediatr Child Health. 2004 Sep-Oct;40(9-10):556-8. doi: 10.1111/j.1440-1754.2004.00463.x. PMID 15367152
- [Background] Starreveld E, Starreveld AA. Status epilepticus. Current concepts and management. Can Fam Physician. 2000 Sep;46:1817-23. PMID 11013800
- [Background] Scheepers M, Scheepers B, Clarke M, Comish S, Ibitoye M. Is intranasal midazolam an effective rescue medication in adolescents and adults with severe epilepsy? Seizure. 2000 Sep;9(6):417-22. doi: 10.1053/seiz.2000.0425. PMID 10985999
- [Background] Jeannet PY, Roulet E, Maeder-Ingvar M, Gehri M, Jutzi A, Deonna T. Home and hospital treatment of acute seizures in children with nasal midazolam. Eur J Paediatr Neurol. 1999;3(2):73-7. doi: 10.1053/ejpn.1999.0185. PMID 10700542
- [Background] Treatment of convulsive status epilepticus. Recommendations of the Epilepsy Foundation of America's Working Group on Status Epilepticus. JAMA. 1993 Aug 18;270(7):854-9. PMID 8340986
- [Background] Chamberlain JM, Altieri MA, Futterman C, Young GM, Ochsenschlager DW, Waisman Y. A prospective, randomized study comparing intramuscular midazolam with intravenous diazepam for the treatment of seizures in children. Pediatr Emerg Care. 1997 Apr;13(2):92-4. doi: 10.1097/00006565-199704000-00002. PMID 9127414
- [Background] Fisgin T, Gurer Y, Senbil N, Tezic T, Zorlu P, Okuyaz C, Akgun D. Nasal midazolam effects on childhood acute seizures. J Child Neurol. 2000 Dec;15(12):833-5. doi: 10.1177/088307380001501219. PMID 11198507
- [Background] Fisgin T, Gurer Y, Tezic T, Senbil N, Zorlu P, Okuyaz C, Akgun D. Effects of intranasal midazolam and rectal diazepam on acute convulsions in children: prospective randomized study. J Child Neurol. 2002 Feb;17(2):123-6. doi: 10.1177/088307380201700206. PMID 11952072
- [Background] Kutlu NO, Yakinci C, Dogrul M, Durmaz Y. Intranasal midazolam for prolonged convulsive seizures. Brain Dev. 2000 Sep;22(6):359-61. doi: 10.1016/s0387-7604(00)00155-8. PMID 11042416
- [Background] Lahat E, Goldman M, Barr J, Bistritzer T, Berkovitch M. Comparison of intranasal midazolam with intravenous diazepam for treating febrile seizures in children: prospective randomised study. BMJ. 2000 Jul 8;321(7253):83-6. doi: 10.1136/bmj.321.7253.83. PMID 10884257
- [Background] Lahat E, Goldman M, Barr J, Bistritzer T, Berkovitch M. Intranasal midazolam as a treatment of autonomic crisis in patients with familial dysautonomia. Pediatr Neurol. 2000 Jan;22(1):19-22. doi: 10.1016/s0887-8994(99)00109-5. PMID 10669200
- [Background] Lahat E, Goldman M, Barr J, Eshel G, Berkovitch M. Intranasal midazolam for childhood seizures. Lancet. 1998 Aug 22;352(9128):620. doi: 10.1016/S0140-6736(05)79574-X. No abstract available. PMID 9746026
- [Background] Lahat E. A prospective, randomized study comparing intramuscular midazolam with intravenous diazepam for the treatment of seizures in children. Pediatr Emerg Care. 1997 Dec;13(6):449. No abstract available. PMID 9435015
- [Background] McGlone R, Smith M. Intranasal midazolam. An alternative in childhood seizures. Emerg Med J. 2001 May;18(3):234. doi: 10.1136/emj.18.3.234. No abstract available. PMID 11354231
- [Background] Rainbow J, Browne GJ, Lam LT. Controlling seizures in the prehospital setting: diazepam or midazolam? J Paediatr Child Health. 2002 Dec;38(6):582-6. doi: 10.1046/j.1440-1754.2002.00046.x. PMID 12410871
- [Background] Scott RC, Besag FM, Neville BG. Buccal midazolam and rectal diazepam for treatment of prolonged seizures in childhood and adolescence: a randomised trial. Lancet. 1999 Feb 20;353(9153):623-6. doi: 10.1016/S0140-6736(98)06425-3. PMID 10030327
- [Background] Wallace SJ. Nasal benzodiazepines for management of acute childhood seizures? Lancet. 1997 Jan 25;349(9047):222. doi: 10.1016/S0140-6736(05)64856-8. No abstract available. PMID 9014904
- [Background] Wroblewski BA, Joseph AB. The use of intramuscular midazolam for acute seizure cessation or behavioral emergencies in patients with traumatic brain injury. Clin Neuropharmacol. 1992 Feb;15(1):44-9. doi: 10.1097/00002826-199202000-00006. PMID 1576597
- [Background] Pellock JM. Status epilepticus in children: update and review. J Child Neurol. 1994 Oct;9 Suppl 2:27-35. PMID 7806783
- [Background] Verity CM. Do seizures damage the brain? The epidemiological evidence. Arch Dis Child. 1998 Jan;78(1):78-84. doi: 10.1136/adc.78.1.78. No abstract available. PMID 9534684
- [Background] Alldredge BK, Wall DB, Ferriero DM. Effect of prehospital treatment on the outcome of status epilepticus in children. Pediatr Neurol. 1995 Apr;12(3):213-6. doi: 10.1016/0887-8994(95)00044-g. PMID 7619187
- [Background] Knoester PD, Jonker DM, Van Der Hoeven RT, Vermeij TA, Edelbroek PM, Brekelmans GJ, de Haan GJ. Pharmacokinetics and pharmacodynamics of midazolam administered as a concentrated intranasal spray. A study in healthy volunteers. Br J Clin Pharmacol. 2002 May;53(5):501-7. doi: 10.1046/j.1365-2125.2002.01588.x. PMID 11994056
- [Background] Mahmoudian T, Zadeh MM. Comparison of intranasal midazolam with intravenous diazepam for treating acute seizures in children. Epilepsy Behav. 2004 Apr;5(2):253-5. doi: 10.1016/j.yebeh.2004.01.003. PMID 15123028
- [Background] Vilke GM, Sharieff GQ, Marino A, Gerhart AE, Chan TC. Midazolam for the treatment of out-of-hospital pediatric seizures. Prehosp Emerg Care. 2002 Apr-Jun;6(2):215-7. doi: 10.1080/10903120290938571. PMID 11962570
- [Derived] Holsti M, Dudley N, Schunk J, Adelgais K, Greenberg R, Olsen C, Healy A, Firth S, Filloux F. Intranasal midazolam vs rectal diazepam for the home treatment of acute seizures in pediatric patients with epilepsy. Arch Pediatr Adolesc Med. 2010 Aug;164(8):747-53. doi: 10.1001/archpediatrics.2010.130. PMID 20679166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from a pediatric Neurology clinic.
Groups:
- Intranasal Midazolam: 0.2 mg/kg Intranasal Midazolam for a seizure longer than 5 minutes
- Rectal Diazepam: 0.3-0.5 Rectal Diazepam for a seizure lasting longer than 5 minutes
Period: Overall Study
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Started | 179 | 179
Completed | 50 | 42
Not Completed | 129 | 137
Not completed — They did not have a seizure requiring tx | 129 | 137

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Midazolam | Rectal Diazepam | Total
Number analyzed (Participants) | 50 | 42 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 42 | 92
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6.8 (5.0) | 7.3 (4.5) | 7.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 50 | 42 | 92

OUTCOME MEASURES:

1. Primary Outcome: Length of Seizure After Study Medication Administration
Description: Length of seizure.
Time Frame: 24 hours
Population: Analysis was per protocol
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Intranasal Midazolam; Rectal Diazepam: Median time to seizure cessation from medication administration to seizures stop time.
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
Minutes | 3.0 (15.7) [1 to 10] | 4.3 (11.3) [2 to 14.5]

2. Secondary Outcome: Respiratory Depression Requiring Intubation
Description: Respiratory depression was defined as intubation at Emergency Department discharge.
Time Frame: 24 hours
Population: Analysis was per protocol
Measure: Number; unit: participants
Groups:
- Intranasal Midazolam: Patients who required oxygen at discharge from the Emergency Department
- Rectal Diazepam: Includes intubation
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 1 [0.0 to 8.3] | 0 [0 to 5]
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 0.8

3. Secondary Outcome: Number of Patients Who Needed Additional Medication to Treat the Seizure in the Emergency Department Within 24 Hours
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 5 [2 to 12] | 5 [4 to 15]
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI [0.2 to 3.9]

4. Secondary Outcome: Number of Patients Needed to be Seen or Treated in the Emergency Department for Their Seizure and Use of Study Medication.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 21 | 17
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 1.1, 95% CI [0.4 to 2.7]

5. Secondary Outcome: Number of Patients That Were Admitted to the Hospital After Their Seizure and Use of Study Medication.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 4 [1 to 10] | 3 [1 to 8]
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 1.1, 95% CI [0.2 to 8.2]

6. Secondary Outcome: Number of Patients Who Had a Repeat Seizure Within 12 Hours After Their Seizure Who Used Study Medication
Time Frame: 12 hours
Measure: Number; unit: participants
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 1 [0 to 5] | 1 [0 to 5]
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI [0.0 to 67.3]

7. Secondary Outcome: Respiratory Depression Requiring Oxygen at Discharge From the Emergency Department.
Description: Respiratory depression was defined as requiring oxygen at discharge from the Emergency Department.
Time Frame: 24 hours
Population: Analysis was per protocol
Measure: Number; unit: participants
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Number analyzed (Participants) | 50 | 42
participants | 3 | 1
Statistical Analysis 1: Comparison: Intranasal Midazolam vs Rectal Diazepam; Test type: Superiority or Other; Odds Ratio (OR) = 2.6, 95% CI [0.2 to 140.7]

ADVERSE EVENTS:
Arm/Group | Intranasal Midazolam | Rectal Diazepam
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/42
Other Adverse Events (participants affected / at risk) | 0/50 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Midazolam (N=50) | Rectal Diazepam (N=42)
Intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No